CLINICAL TRIAL: NCT06323746
Title: Exploring Heart Rate Variability, EEG Pattern, and Corticomuscular Coherence After Cervical Sagittal Alignment Restoration: A Randomized Controlled Trial Investigation
Brief Title: Exploring Heart Rate Variability, EEG Pattern, and Corticomuscular Coherence After Cervical Sagittal Alignment Restoration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Professor and Chairman of Physiotherapy, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR-EEG-CSAR
Record Dates: First submitted 2024-03-01; First posted 2024-03-21 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cervical Lordosis
Keywords: Cervical Lordosis; Athlete; Electroencephalography; Heart Rate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Permuted block randomization to ensure an equal number of allocations in each of the two groups (intervention and wait list group). Each random block will be stored in opaque sealed envelopes consecutively numbered with a third researcher. Once each participant officially joins the study the researcher will open the subsequent envelop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denneroll Group (Experimental): The participants will be instructed to lie flat on their back on the ground with their legs extended and arms by their sides and gently folded across their stomach. The subject will place the Denneroll on the ground and the examiner positions the apex of the Denneroll.
  The apex of the Denneroll orthotic will be placed in one of three regions based on lateral cervical radiographic displacements.
  Interventions: Device: Denneroll cervical traction orthodontic
- Wait List (Other): This group will receive the same posture correction program after all data will be collected.
  Interventions: Device: Denneroll cervical traction orthodontic

INTERVENTIONS:
Device: Denneroll cervical traction orthodontic — The duration of each session will start at approximately three minutes and increase by one minute per session until reaching the goal of 20 minutes per session. The intervention will be repeated three times per week for 10 weeks in the supervised setting.

SUMMARY:
The goal of this Randomized clinical trial is to learn about how fixing neck curvature and head posture right away affects heart rate, brainwaves, and muscle coordination in college athletes. The main question it aims to answer:

- Whether forward head posture (FHP) may play a crucial role in affecting heart rate variability, brainwaves, and muscle coordination.

DETAILED DESCRIPTION:
Background: Restoring normal cervical spine alignment has emerged as one of the most important clinical outcomes in healthcare. However, the question of whether cervical biomechanical dysfunction manifesting as forward head posture (FHP) may play a crucial role in affecting heart rate variability, as an indicator of the autonomic nervous system, electroencephalography (EEG) pattern, as indictor for brain waves, and corticomuscular coherence, as an indicator of the functional connection between the cortex and muscles during continuous muscle contractions among collegiate athletes has not been answered yet.

Objective: To investigate the immediate and long-term effects of cervical lordosis restoration and forward head correction using the Denneroll™ on heart rate variability, EEG pattern, and corticomuscular coherence among collegiate athletes.

Methods: Eighty asymptomatic subjects with a definite hypolordotic cervical spine and FHP will be randomly assigned to an experimental group or a control group. The experimental group will receive the Denneroll™ cervical traction while the control group will be considered as a wait list to start the intervention after completion of the experimental group. Interventions will be applied 3 times per week for a period of 10 weeks. Changes in heart rate variability, EEG pattern and corticomuscular coherence will be assessed at three-time intervals: at baseline, after 10 weeks of intervention, and at 6-months follow up with no further interventions.

ELIGIBILITY:
Inclusion Criteria:

* Anterior head translation (AHT) >15 mm
* Absolute rotatory angle C2 to C7 is <25°
* Athletic student

Exclusion Criteria:

* Inflammatory joint disease or other systemic pathologies
* Prior history of overt injury and surgery relating to the musculoskeletal system, or disorder related to the spine and extremities
* Musculoskeletal pain in the previous three months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cervical Sagittal Alignment Radiographs | Baseline (pre-treatment), week 10 (upon completion) and after 6 months
  The change of cervical lordosis from the absolute rotatory angle C2-7.
Cervical Sagittal Alignment Radiographs | Baseline (pre-treatment), week 10 (upon completion) and after 6 months
  The amount of the change in the anterior head translation from the horizontal offset of the posterior superior body corner of C2 relative to the vertical line.

SECONDARY OUTCOMES:
Heart rate Variability (HRV) physiological parameter | Baseline (pre-treatment), week 10 (upon completion) and after 6 months
  The change in Heart rate through Electrocardiographic recordings (ECG) will be monitored using a Nexus-10 physiologic monitoring system. Recordings will be made simultaneously through three separate channels. The ground electrode will be placed below the left clavicle, the cathode (-) below the right clavicle and the anode (+) will be placed on the third rib, in line with the ground.
  HRV time parameter will be calculated from respiratory rate (RR) intervals (Standard deviation of the normal to normal intervals (SDNN), Root-mean-square of the successive normal sinus RR interval difference (RMSSD) and the percentage of absolute differences between successive normal RR intervals that exceed 50 ms (pNN50)).
  HRV frequency domain variable will include total power, high frequency (HF) and low frequency (LF) power (measured in ms2) and LF:HF ratio were derived from spectral analysis of successive R-R intervals.
Corticomuscular Coherence | Baseline (pre-treatment), week 10 (upon completion) and after 6 months
  The change in the ratio between Muscle activity through Electromyography (EMG) and brain waves through Electroencephalograph (EEG)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.